CLINICAL TRIAL: NCT04979936
Title: Early Laparoscopic Cholecystectomy Versus Percutaneous Cholecystostomy Followed by Delayed Laparoscopic Cholecystectomy in Patients With Grade II Acute Cholecystitis According to Tokyo Guidelines
Brief Title: Early Laparoscopic Cholecystectomy Versus Percutaneous Cholecystostomy in Grade II Acute Cholecystitis Guidelines
Acronym: PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/11
Record Dates: First submitted 2021-07-17; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Acute Cholecystitis; Empyema, Gallbladder
Keywords: moderate acute cholecystitis, percutaneous cholecystostomy
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early laparoscopic cholecystectomy (Active Comparator): early laparoscopic cholecystectomy
  Interventions: Procedure: laparoscopic cholecystectomy
- percutaneous cholecystostomy (Active Comparator): percutaneous cholecystostomy first followed by delayed laparoscopic cholecystectomy
  Interventions: Procedure: percutaneous cholecystostomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy
  Arms: early laparoscopic cholecystectomy
Procedure: percutaneous cholecystostomy
  Arms: percutaneous cholecystostomy

SUMMARY:
The aim of this study is to compare between early laparoscopic cholecystectomy versus percutaneous cholecystostomy followed by delayed interval laparoscopic cholecystectomy as regards the operative and postoperative complications

DETAILED DESCRIPTION:
A-Study setting: Department of Surgery, main university hospital, Faculty of Medicine, Alexandria University, Egypt. The study was approved by the Ethics Committee of our institution.

B-Study design: Retrospective clinical trial C-Study subjects: The target population are patients with preoperative diagnosis of grade II acute cholecystitis Those patients were subjected to surgery either early laparoscopic cholecystectomy or delayed laparoscopic cholecystectomy after percutaneous cholecystostomy

Inclusion criteria of the study patients:

-Specific written informed consent approved by our Institution's Ethics Committee was obtained from all the treated patients.

Exclusion criteria:

-contraindication to laparoscopy,Refusal of study participation, cirrhosis, grade I or III acute cholecystitis D-Sample size calculation: a minimum sample size required per group is 88 to detect decline in the proportion of the primary outcome from 20% to 5%, at 5% level of significance and 80% power.

E-Sampling technique: By using eligibility criteria, 220 patients that were planned to undergo laparoscopic Cholecystectomy were randomly selected from the surgery department in main university hospital, Faculty of Medicine, Alexandria University. They were randomly separated into two groups:

An experiment group: (90 patients) underwent percutaneous cholecystostomy followed by delayed interval laparoscopic cholecystectomy A control group: (130 patients) underwent early laparoscopic cholecystectomy. All the participants were initially evaluated and re-evaluated during follow up period of 30 days for the outcome measures. Non blinded trial was done due to difficulty in using blinding in operative intervention.

Methods: every patient in the study sample was subjected to the followings:

1. History
2. Examination:
3. Investigations ( pre and postoperative):

   Laboratory: WBC, CRP, lever functions Radiologic imaging: ultrasonography, CT abdomen
4. Intervention: An experiment group: underwent percutaneous cholecystostomy followed by delayed interval laparoscopic cholecystectomy.

   A control group: underwent early laparoscopic cholecystectomy.

   Surgical Technique: laparoscopic cholecysctomy Postoperative Course: post-operative complications
5. Outcome Measurement and Follow-Up

   * Follow up period: both groups were re-evaluated at 1, 2, 6 months. They were evaluated for the positive and negative outcome measures. There were no cases lost to follow up.
   * Outcome measures that were assessed after the follow up period were:
   * Primary outcome measures: operative and postoperative complications as conversion, biliary injury, bowel injury, they were assessed by clavien dindo classification
   * Secondary Outcome measures: ASA score, Tokyo score and some investigations.

Statistical analysis Statistical analysis was performed using the Statistical Package for the Social Sciences (SPSS) version 20 software (SPSS, Inc., Chicago, IL, USA). Quantitative variables were summarized using mean and standard deviation after data exploration using the Kolmogorov- Smirnov test. Qualitative variables were described using number and percent. Associations between the two groups and other categorical variables were assessed using Chi-square test (Fisher or Monte Carlo). Comparisons between the two groups as regards the quantitative variables were assessed using Student t-test. All Statistical tests were done at 5% level of Significance.

Risk estimates were calculated as Relative risk, Absolute risk reduction, Number needed to treat and population Attributable Risk percentage to detect the risk of development of the intraoperative and postoperative complications in the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* patients with one of the criteria stated by grade II (moderate) Tokyo guidelines for acute cholecystitis who were managed either by early LC or by a bridging PC followed by delayed LC.

Exclusion Criteria:

* grade I or III acute cholecystitis
* common bile duct stones or jaundice,
* Liver cirrhosis,
* severe upper abdominal adhesions,
* acalculous cholecystitis
* major comorbidities in which laparoscopic surgery is contraindicated.
* those who followed a conservative treatment for acute cholecystitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
operative difficulties as conversion, operative time, biliary injury | at the time of cholecysctomy
  as assessed by the main surgeon
postoperative complications | 30 days after the operation
  as assessed by clavien dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: HANY MK EL-HADDAD, professor, Principal Investigator — alexandria university, faculty of medicine
Locations (2):
- Egypt (2):
  - Alexandria university, Alexandria
  - Faculty of Medicine, Alexandria

IPD SHARING:
Plan to Share IPD: No
data extracted from the hospital records. it is difficult to bring these data into public